CLINICAL TRIAL: NCT04186468
Title: Piloting an ICU Follow-up Clinic to Improve Health Related Quality of Life After a Prolonged Intensive Care Stay
Brief Title: ICU Follow-up After Prolonged Intensive Care Stay
Acronym: PINA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Otto-von-Guericke University Magdeburg (Other)
Collaborators: University of Regensburg (Other); University Hospital Regensburg (Other)
Responsible Party: Principal Investigator, Christian J. Apfelbacher, Director, Institute of Social Medicine and Health Systems Research, Otto-von-Guericke University Magdeburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PINA-2019; VF_2016-076 (Other: Federal Joint Committee (G-BA) application); 01VSF16056 (Other Grant/Funding Number: Innovation Fund of the Federal Joint Committee (G-BA)); 19-1522-101 (Other: Ethics Committee, University of Regensburg)
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Critical Illness; PICS; Post Intensive Care Syndrome
Keywords: PICS; ICU; Intensive Care Unit; Post Intensive Care Syndrome; Follow-up clinic; Intensive care unit-acquired weakness; Critical illness polyneuropathy; Health-related quality of life; Critical care; Muscle weakness
MeSH Terms: conditions — Critical Illness; postintensive care syndrome; Polyneuropathies; Muscle Weakness

STUDY DESIGN:
Intervention Model Description: The treatment group will supported by activities of an ICU follow-up clinic. The control group will receive usual care.
Who Masked: Outcomes Assessor
Masking Description: Group allocation will be masked during analysis of the primary outcome. Masking and unmasking will be done by a Trust Center by coding both groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICU follow-up clinic (Experimental): Participants will be invited to visit the ICU follow-up clinic.
  Interventions: Other: ICU follow-up clinic
- Usual care (No Intervention): Participants will solely receive usual care.

INTERVENTIONS:
Other: ICU follow-up clinic — The intervention aims at improving health-related quality of life and will contain three components: information, consultation and networking. More information will be available for the participants from the intensive care stay onwards, e.g. an information brochure, and during the entire follow-up period, e.g. by contacting the outpatient clinic via telephone. Participants will be invited to visit the ICU follow-up clinic at least once during the first six months after discharge from ICU. During the visits, participants will be screened for symptoms of PICS and, if required, referred to specialists for further treatment. The aim of the networking part is to improve the exchange between the health sectors and disciplines, e.g. through a special referral letter from the ICU follow-up clinic, and thus to provide a network of outpatient care providers for the former ICU patients.
  Arms: ICU follow-up clinic

SUMMARY:
Treatment in the intensive care unit (ICU) for more than five days often leads to chronic physical, cognitive and psychological complaints, such as post-traumatic stress disorders, muscle weakness, depression, anxiety and adjustment disorders. This is referred to as Post Intensive Care Syndrome (PICS). So far, there have been only a few studies investigating this syndrome.

The aim of this pilot study is to test the effectiveness and feasibility of an ICU follow-up clinic, which our study team developed in a participatory process involving patients, caregivers, health care providers and researcher.

For this purpose, the participants will be randomly assigned to a group with treatment in this follow-up clinic or to a group with usual care. Both groups will then be compared.

DETAILED DESCRIPTION:
Intensive care unit (ICU) survivors often suffer from cognitive, physical and psychological impairments, known as Post Intensive Care Syndrome (PICS). In order to improve healthcare of these patients in general and medical follow-up in particular, various aftercare models have been developed in different countries, including ICU follow-up clinics. So far, there is no uniform concept for an ICU follow-up clinic. Therefore, there is insufficient evidence whether or which concept of an ICU follow-up clinic is effective in addressing the health needs of ICU survivors. Within our study "Piloting an ICU Follow-up Clinic to Improve Health Related Quality of Life After a Prolonged Intensive Care Stay" (German abbreviation PINA), a concept for an ICU follow-up clinic was developed and will be tested in a pilot randomized controlled trial (RCT).

The study design comprises a pilot RCT with intervention and control (usual care) arms and an additional qualitative and quantitative process evaluation. One hundred ICU patients (fifty per arm) of three ICUs at University Hospital Regensburg will be enrolled as participants. Potential participants have to be older than eighteen years with an ICU stay of at least five days, a SOFA (sequential organ failure assessment) score greater than five and a life expectancy of more than six months.

The intervention aims at improving health-related quality of life and will contain three components: information, consultation and networking. More information (e.g. about sequelae after ICU, treatment options) will be available for the participants from the intensive care stay onwards, e.g. an information brochure, and during the entire follow-up period, e.g. by contacting the ICU follow-up clinic via telephone. Participants will be invited to visit the ICU follow-up clinic at least once during the first six months after discharge from ICU. During the visits, participants will be screened for symptoms of PICS and, if required, referred to specialists for further treatment. The aim of the networking part is to improve the exchange between the health sectors and disciplines involved in the treatment of the patients, e.g. through a special referral letter from the ICU follow-up clinic, and thus to provide a network of outpatient care providers for the former ICU patients.

Efficacy Outcomes: Health-related quality of life (HRQOL) will be assessed as primary outcome by the Short-Form-12 Questionnaire (SF-12). As secondary outcomes patient-reported outcomes regarding physical, psychological and social functioning are assessed. Additionally, HRQOL of next of kin is assessed. All outcomes are assessed at six months after discharge from ICU. Feasibility Outcomes: Qualitative and quantitative evaluation will be used for exploring reasons for non-participation and the intervention's acceptability to patients, caregivers and health care providers The PINA study will determine feasibility and efficacy of a complex intervention in a pilot RCT to enhance follow-up care of ICU survivors. The pilot study is an important step for further studies in the field of ICU aftercare and especially for the implementation of a pragmatic multicenter RCT.

ELIGIBILITY:
Inclusion Criteria:

* duration of ICU stay more than five days
* sequential organ failure assessment score (SOFA) greater than five
* expected survival time greater than six months
* written informed consent

Exclusion Criteria:

* minor participants under the age of eighteen
* no written informed consent (unable or unwilling)
* unable to complete questionnaires
* insufficient German language skills

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Health related quality of life, physical component summary score (HRQOL-PCS) | Six months after ICU discharge
  HRQOL will be assessed six months after discharge from the intensive care unit (ICU) by the Short Form-12 self-report questionnaire (SF-12) physical component summary score (PCS) (Ware, 1996). The German translation (Bullinger, 1998) will be used. Scores can range between zero and one hundred, with higher values indicating higher HRQOL.

SECONDARY OUTCOMES:
Health related quality of life, mental component summary score (HRQOL-MCS) | Six months after ICU discharge
  HRQOL will be assessed six months after discharge from the intensive care unit (ICU) by the Short Form-12 self-report questionnaire (SF-12) mental component summary score (MCS) (Ware, 1996). The German translation (Bullinger, 1998) will be used. Scores can range between zero and one hundred, with higher values indicating higher HRQOL.
Activities of Daily Living (ADL) | Six months after ICU discharge
  ADL will be assessed by the Barthel-Index (Mahoney, 1965) in German translation (Lübke, 2004), which evaluates ten everyday functions. The degree of independence or care dependence can be assessed on a score ranging between zero (complete need for care) and one hundred points (independence).
Chair Rise Test | Six months after ICU discharge
  The Chair Rise Test (Cooper, 2010 and Fuchs, 2013) will be used to assess participants' physical functioning. Anyone who cannot get up from a chair at normal height five times in a row in eleven seconds or less without supporting himself with his arms is considered to be at risk of falling.
Hand Grip Strength | Six months after ICU discharge
  As an indicator for the general muscular strength (Beaton, 1995, Bobos, 2019), we will measure the hand grip strength with a dynamometer (Jamar Plus+ Digital Hand Dynamometer). Values can range fron zero to ninety kilogram, whereby higher values indicate a higher gripping force.
Post-Traumatic Stress Syndrome 10-Questions Inventory (PTSS-10) | Six months after ICU discharge
  The PTSS-10 (Weisæth, 1989) will be used in the German translation (Maercker, 1998) to assess participants' risk of post traumatic stress disorders. Each symptom is rated from one (never) to seven (always). A total score of more than thirty-five predicts a likely diagnosis of post-traumatic stress disorder (PTSD).
Short Form German Patient Health Questionnaire (PHQ-D) | Six months after ICU discharge
  The PRIME MD Brief Patient Health Questionnaire, PHQ (Spitzer, 1999) will be used in the German short form translation PHQ-D (Loewe, 2002) to assess psychopathological symptoms (anxiety, panic disorder or depression). Score values can range from zero to twenty-seven, with higher values being a good indicator for psychiatric diagnoses.
Inpatient and outpatient health care utilization. | Six months after ICU discharge
  The extent of ambulatory and stationary health care use among the former ICU patients will be assessed by self-reported contacts with health services using a questionnaire as a proxy for morbidity. These contacts can range from zero to unlimited. A higher level of contacts indicates a weaker state of health.
Health related quality of life (HRQOL) of next of kin | Six months after ICU discharge of the participant
  HRQOL of next of kin will be assessed also six months after discharge of the participant by the Short Form-12 self-report questionnaire (SF-12) PCS and MCS (Ware, 1996) after informed consent was obtained from the the respective relative. The German translation (Bullinger, 1998) will be used. Scores of both component scales can range between zero and one hundred, with higher values indicating higher HRQOL.

CONTACTS AND LOCATIONS:
Overall Officials: Christian J Apfelbacher, Prof.Dr.PhD, Principal Investigator — Otto-von-Guericke University Magdeburg
Locations (3):
- Germany (3):
  - Institute of Social Medicine and Health Systems Research, Magdeburg
  - Department for Epidemiology and Preventive Medicine, Regensburg
  - University Hospital, Regensburg

REFERENCES:
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] MAHONEY FI, BARTHEL DW. FUNCTIONAL EVALUATION: THE BARTHEL INDEX. Md State Med J. 1965 Feb;14:61-5. No abstract available. PMID 14258950
- [Background] Fuchs J, Busch MA, Gosswald A, Holling H, Kuhnert R, Scheidt-Nave C. [Physical and cognitive capabilities among persons aged 65-79 years in Germany: results of the German Health Interview and Examination Survey for Adults (DEGS1)]. Bundesgesundheitsblatt Gesundheitsforschung Gesundheitsschutz. 2013 May;56(5-6):723-32. doi: 10.1007/s00103-013-1684-7. German. PMID 23703491
- [Background] Cooper R, Kuh D, Cooper C, Gale CR, Lawlor DA, Matthews F, Hardy R; FALCon and HALCyon Study Teams. Objective measures of physical capability and subsequent health: a systematic review. Age Ageing. 2011 Jan;40(1):14-23. doi: 10.1093/ageing/afq117. Epub 2010 Sep 15. PMID 20843964
- [Background] Weisaeth L. Torture of a Norwegian ship's crew. The torture, stress reactions and psychiatric after-effects. Acta Psychiatr Scand Suppl. 1989;355:63-72. PMID 2624136
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] Beaton DE, O'Driscoll SW, Richards RR. Grip strength testing using the BTE work simulator and the Jamar dynamometer: a comparative study. Baltimore Therapeutic Equipment. J Hand Surg Am. 1995 Mar;20(2):293-8. doi: 10.1016/s0363-5023(05)80029-2. PMID 7775773
- [Background] Bobos P, Nazari G, Lu Z, MacDermid JC. Measurement Properties of the Hand Grip Strength Assessment: A Systematic Review With Meta-analysis. Arch Phys Med Rehabil. 2020 Mar;101(3):553-565. doi: 10.1016/j.apmr.2019.10.183. Epub 2019 Nov 13. PMID 31730754
- [Background] Bullinger M, Kirchberger I. Der SF-36 Fragebogen zum Gesundheitszustand (SF-36). Handbuch für die deutschsprachige Fragebogenversion Göttingen, Hogrefe, 1998.
- [Background] Löwe B, Spitzer R, Zipfel S, Herzog W. PHQ-D Gesundheitsfragebogen für Patienten (German Version of the Patient Health Questionnaire). Karlsruhe: Pfizer, 2002.
- [Background] Maercker, A. Posttraumatische Stress Skala-10 (PTSS-10) - deutsche Version modifiziert nach Schüffel u. Schade. Unveröffentlichtes Manuskript, Universität Zürich, Klinische Psychologie II, 1998.
- [Background] Lubke N, Meinck M, Von Renteln-Kruse W. [The Barthel Index in geriatrics. A context analysis for the Hamburg Classification Manual]. Z Gerontol Geriatr. 2004 Aug;37(4):316-26. doi: 10.1007/s00391-004-0233-2. German. PMID 15338161
- [Derived] Drewitz KP, Hasenpusch C, Bernardi C, Brandstetter S, Fisser C, Pielmeier K, Rohr M, Brunnthaler V, Schmidt K, Malfertheiner MV, Apfelbacher CJ. Piloting an ICU follow-up clinic to improve health-related quality of life in ICU survivors after a prolonged intensive care stay (PINA): feasibility of a pragmatic randomised controlled trial. BMC Anesthesiol. 2023 Oct 14;23(1):344. doi: 10.1186/s12871-023-02255-1. PMID 37838669
- [Derived] Rohr M, Brandstetter S, Bernardi C, Fisser C, Drewitz KP, Brunnthaler V, Schmidt K, Malfertheiner MV, Apfelbacher CJ. Piloting an ICU follow-up clinic to improve health-related quality of life in ICU survivors after a prolonged intensive care stay (PINA): study protocol for a pilot randomised controlled trial. Pilot Feasibility Stud. 2021 Mar 30;7(1):90. doi: 10.1186/s40814-021-00796-1. PMID 33785064